CLINICAL TRIAL: NCT00707538
Title: A Phase I Dosimetry, Biodistribution and Safety Study of BMS747158 in Healthy Subjects Undergoing 2-Day Rest/Stress Positron Emission Tomography
Brief Title: A Phase I Study in Healthy Volunteers to Assess Dosimetry and Safety Following Injection of BMS747158 at Stress
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Lantheus Medical Imaging (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: BMS747158-102
Record Dates: First submitted 2008-06-27; First posted 2008-07-01 (Estimated); Last update posted 2020-11-10 (Actual); Status verified 2011-08

CONDITIONS: Healthy Volunteers
MeSH Terms: interventions — BMS 747158-02

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 1 (Experimental)
  Interventions: Drug: BMS747158

INTERVENTIONS:
Drug: BMS747158 — 2 IV injection of ~11 mCi (total) F-18 labeled compound

SUMMARY:
The purpose of this clinical research study is to learn the biodistribution of injection of BMS747158 at stress and assess the safety of two doses of BMS747158

ELIGIBILITY:
Inclusion Criteria:

* age 18-40
* BMI 18-30 kg/m2
* No active or chronic illnesses
* If female: not pregnant, use of birth control or not of child-bearing potential

Exclusion Criteria:

* Significant active or chronic illness
* Any neurological disorder
* GI disease within 3 months
* Recent infection
* Major surgery within 4 weeks
* Donation of blood within 4 weeks
* Blood transfusion within 4 weeks
* Recent history drug/alcohol abuse
* Head trauma
* Significant screening ECG, EEG, lab tests, physical exam and vital signs abnormalities
* Prescription or OTC drugs within 2 weeks
* Exposure to any other investigational

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2008-06; Primary Completion 2008-10 (Actual); Study Completion 2008-10 (Actual)

PRIMARY OUTCOMES:
Dosimetry analysis following whole body imaging after stress injection | Imaging takes place approximately 0 - 300 minutes post injection

SECONDARY OUTCOMES:
Safety analysis following vital signs, ECGs, EEG, neuro and physical exams, telephone and visit follow up, and blood draws for chemistry and hematology post injection of BMS747158 at rest and stress | Screening (14 days prior to dosing) through 14 days post dose administration

CONTACTS AND LOCATIONS:
Overall Officials: Jamshid Maddahi, MD, Principal Investigator — University of California, Los Angeles
Locations (2):
- United States (2):
  - UCLA Medical Center, Los Angeles, California
  - John Hopkins University, Baltimore, Maryland